CLINICAL TRIAL: NCT03163017
Title: Does Intraoperative 3D Fluoroscopy Accurately Assess Syndesmotic Reduction Following Traumatic Ankle Injury?
Brief Title: Assessment of Ability of 3D Fluorscopy in Aiding Accurate Syndesmotic Reduction Following Traumatic Ankle Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: AO Trauma North America (Unknown)
Responsible Party: Principal Investigator, Joshua L Gary, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0840
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Displaced Ankle Fractures
Keywords: 3D Fluoroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 2D Fluoroscopy then 3D Fluoroscopy (Experimental): Patients with syndesmotic instability will undergo reduction of the syndesmosis followed by provisional fixation with a clamp or Kirshner wire. The reduction quality will be initially compared to the contralateral ankle mortise and talar-dome lateral radiographs using the technique of Summers et al (2D Fluoroscopy). After the attending surgeon is satisfied with the reduction quality, 3D fluoroscopy will be used to generate additional images to assess syndesmotic and fibular reductions. Both 2D and 3D Fluoroscopy will be performed using device "Ziehm Vision RFD 3D image-intensified fluoroscopic x-ray system".
  Interventions: Device: 2D Fluoroscopy; Device: 3D Fluoroscopy

INTERVENTIONS:
Device: 2D Fluoroscopy — Patients with syndesmotic instability will undergo reduction of the syndesmosis followed by provisional fixation with a clamp or Kirshner wire. The reduction quality will be initially compared to the contralateral ankle mortise and talar-dome lateral radiographs using the technique of Summers et al i.e. 2D Fluoroscopy using device Ziehm Vision RFD 3D image-intensified fluoroscopic x-ray system.
Device: 3D Fluoroscopy — After the attending surgeon is satisfied with the reduction quality from 2D Fluoroscopy, 3D fluoroscopy using device Ziehm Vision RFD 3D image-intensified fluoroscopic x-ray system will be used to generate additional images to assess syndesmotic and fibular reductions.

SUMMARY:
The purpose of this study is to determine if use of new imaging technology termed "3D fluoroscopy" will lead the surgeon to change the position of the fractured bones to a more accurate position.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Patients with unilateral, acute, displaced ankle fractures with preoperative evidence of syndesmotic disruption or intraoperative evidence of syndesmotic instability following malleolar fixation.

Exclusion Criteria:

* Patients skeletally immature;
* Patients less than age 18 years and more than age 75;
* Patients with previous ankle trauma to either ankle;
* Patients with bilateral ankle injuries;
* Patients with previous osseous injuries to the tibia or fibula; and
* Patients with isolated syndesmotic injury and no fracture (i.e. high ankle sprains)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua L Gary, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas at Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 39 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black | 10
  Hispanic | 12
  White | 5
  Unknown | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Which the Surgeon Changed Reduction of Syndesmotic Reduction Because of Information Provided by 3D Fluoroscopy
Description: Patients with syndesmotic instability will undergo reduction of the syndesmosis followed by provisional fixation with a clamp or Kirshner wire. The reduction quality will be initially compared to the contralateral ankle mortise and talar-dome lateral radiographs using the technique of Summers (2D Fluoroscopy). After the attending surgeon is satisfied with the reduction quality, 3D fluoroscopy will be used to generate additional images to assess syndesmotic reductions.
Time Frame: Immediately at the time of 3D Fluoroscopy
Measure: Count of Participants; unit: Participants
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 30
Participants | 14

2. Secondary Outcome: Number of Participants for Which the Surgeon Changed Reduction of Fibular Fracture Reduction Because of Information Provided by 3D Fluoroscopy
Description: Patients with syndesmotic instability will undergo reduction of the syndesmosis followed by provisional fixation with a clamp or Kirshner wire. The reduction quality will be initially compared to the contralateral ankle mortise and talar-dome lateral radiographs using the technique of Summers (2D Fluoroscopy). After the attending surgeon is satisfied with the reduction quality, 3D fluoroscopy will be used to generate additional images to assess fibular fracture reductions.
Time Frame: Immediately at the time of 3D Fluoroscopy
Measure: Count of Participants; unit: Participants
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 30
Participants | 0

3. Secondary Outcome: Pain as Assessed by the AOFAS Score
Description: The patient outcome variables studied will include American Orthopedic Foot and Ankle Society (AOFAS) scores
Time Frame: 3 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

4. Secondary Outcome: Function as Assessed by the AOFAS Score
Description: The patient outcome variables studied will include American Orthopedic Foot and Ankle Society (AOFAS) scores
Time Frame: 3 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

5. Secondary Outcome: Alignment as Assessed by the AOFAS Score
Description: The patient outcome variables studied will include American Orthopedic Foot and Ankle Society (AOFAS) scores
Time Frame: 3 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

6. Secondary Outcome: Pain as Assessed by the AOFAS Score
Description: The patient outcome variables studied will include American Orthopedic Foot and Ankle Society (AOFAS) scores
Time Frame: 6 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

7. Secondary Outcome: Function as Assessed by the AOFAS Score
Description: The patient outcome variables studied will include American Orthopedic Foot and Ankle Society (AOFAS) scores
Time Frame: 6 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

8. Secondary Outcome: Alignment as Assessed by the AOFAS Score
Description: The patient outcome variables studied will include American Orthopedic Foot and Ankle Society (AOFAS) scores
Time Frame: 6 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

9. Secondary Outcome: Pain as Assessed by the PROMIS Score
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) patient physical health outcome measures
Time Frame: 3 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

10. Secondary Outcome: Function as Assessed by the PROMIS Score
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) patient physical health outcome measures
Time Frame: 3 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

11. Secondary Outcome: Pain as Assessed by the PROMIS Score
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) patient physical health outcome measures
Time Frame: 6 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

12. Secondary Outcome: Function as Assessed by the PROMIS Score
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) patient physical health outcome measures
Time Frame: 6 months after 3D Fluoroscopy
Population: Data was not collected for this outcome measure.
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Syndesmotic Malreduction as Assessed by a Single Postoperative Bilateral CT Scan
Description: Malreduction will be determined by comparing uninjured ankle to the injured ankle
Time Frame: 1 day after 3D Fluoroscopy
Measure: Count of Participants; unit: Participants
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
Number analyzed (Participants) | 30
Participants | 3

ADVERSE EVENTS:
Time Frame: Through the time of hospitalization (about 1 day after the procedure)
Arm/Group | 2D Fluoroscopy Then 3D Fluoroscopy
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT03163017/Prot_SAP_000.pdf